CLINICAL TRIAL: NCT04749134
Title: MRI Development for Radiotherapy Planning and Delivery in Non-Patient Volunteers
Acronym: MINION
Status: Recruiting | Type: Observational
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Cynthia Eccles, Head of Radiotherapy Research and Development, The Christie NHS Foundation Trust
Other Study IDs: CFTSp170
Record Dates: First submitted 2021-01-27; First posted 2021-02-11 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Focus of the Study is MRI Sequence Development

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Non-patient volunteers will be scanned on the MR-Linac and MRSIM to facilitate the development, optimisation and validation of MRI protocols at The Christie NHS Foundation Trust.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written consent
* Volunteers must undergo and satisfy MRI safety screening
* Volunteers must be ≥ 16 years of age
* Participants must agree to registration as a non-patient in CWP (the Trust's Electronic Health Record - EHR- system) and have their MRIs read and reported for incidental findings by a clinical radiologist

Exclusion Criteria:

* Any contraindications to MRI identified after MRI safety screening including completion of an MRI Safety Screening Form
* Unable to tolerate MRI scan
* Known Pregnancy
* Known or suspected pathology in body region to be scanned
* Member of study team

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Personnel at The Christie NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Developed and optimised of MRI scanning sequences for use in clinical radiotherapy practice in MR guided radiotherapy | Through study completion - up to 5 years
  on-going development of MRI protocols to be released for clinical use

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie NHS FT, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No